CLINICAL TRIAL: NCT00018031
Title: A Non-Randomized, Open Label, Study to Assess Hepatitis C Viral Kinetics in Predicting the Clinical Response in Patients With Hepatitis C Infection Coinfected With HIV-1 Treated With Peginterferon Alpha-2b and Ribavirin
Brief Title: Peginterferon Alpha-2b And Ribavirin to Treat Hepatitis C in HIV-Infected Patients
Acronym: HEPCPR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Shyamasundaran Kottilil, M.D., Staff Clinician, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 010194; 01-I-0194
Record Dates: First submitted 2001-06-27; First posted 2001-06-28 (Estimated); Results first posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Hepatitis C; HIV Infections
Keywords: Liver Disease; Virologic Response; Immune Mechanisms; Cirrhosis; Eradication; HIV; Hepatitis C
MeSH Terms: conditions — Hepatitis C; HIV Infections; Liver Diseases; Fibrosis | interventions — peginterferon alfa-2b; Ribavirin

ARMS (1):
- 1 (Experimental): Weekly Injection of peginterferon alfa-2b and weight based ribavirin (1-1.2g/day) for 48 weeks
  Interventions: Drug: Peginterferon alfa-2b; Drug: Ribavirin

INTERVENTIONS:
Drug: Peginterferon alfa-2b — Weekly injections for 48 weeks of a dose of 1.5mcg/Kg per week subcutaneously
  Other Names: PegIntron; PEG-Intron; PegIntron Redipen; Sylatron
Drug: Ribavirin — Weight based Ribavirin dosing 1-1.2grams/day in divided (twice daily) doses for a total duration of 48 weeks.
  Other Names: ICN-1229; Copegus; Rebetol; Ribasphere; RBV; RTCA; Rebretron; Ribav; Ribavirine; Tribavirin; Vilona; Viramid; Virazid; Virazole; CAS Number: 36791-04-5

SUMMARY:
This study will evaluate the safety and effectiveness of combination therapy with peginterferon alfa-2b and ribavirin for treating hepatitis C virus (HCV) infection in HIV-infected patients. In studies of patients with hepatitis C alone, interferon alfa-2b plus ribavirin treatment eradicated the HCV in almost half the patients. Peginterferon alfa-2b is a compound that results from attaching a polyethylene glycol molecule to interferon alfa-2b. This compound stays in the blood longer than unmodified interferon alfa-2b, causing a higher blood concentration and thus maintaining activity against the hepatitis C virus.

HIV-infected patients 21 years of age and older with chronic hepatitis C infection and a viral load greater than 2000 copies/mL may be eligible for this 2 1/2-year study. Candidates will be screened with blood and urine tests and possibly a liver biopsy, if a recent one is not available. The liver biopsy is done to determine the severity of liver disease. For this test, patients are admitted to the NIH Clinical Center for 1 to 2 days. A sedative is injected into an arm vein, the skin in the area over the biopsy site is numbed with a local anesthetic, and a needle is inserted rapidly into and out of the liver to obtain a small tissue sample. The patient remains in the hospital overnight for monitoring. A chest X-ray, electrocardiogram (EKG) and liver ultrasound are also done. Within 4 weeks of the screening tests, candidates who appear eligible for the study will have a physical examination, medical history and repeat blood tests. Women who can become pregnant will have serial pregnancy tests throughout the study.

Patients who meet the study criteria and decide to participate will begin treatment with weekly injections under the skin of peginterferon alfa-2b and take ribavirin pills twice a day by mouth. In addition, patients will continue to take all other medications prescribed by their doctor. Clinic visits will be scheduled as follows:

* Days 1, 3, 5, 7, 10 and 21 - Blood will be drawn for safety tests and to measure blood levels of HIV and HCV.
* Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 52, 56 and 64 - Blood and urine tests will be done to determine the side effects of treatment and its effect on the HCV infection.
* Week 48 or end of treatment - Treatment will stop after 48 weeks. At this time, or earlier for those who do not complete the 48 weeks, patients will return to the clinic for a routine test.

DETAILED DESCRIPTION:
Hepatitis C infection occurs in one-third of all HIV-infected individuals. Liver disease has become more clinically significant among patients coinfected with HIV and HCV. Several studies have shown that coinfected individuals develop earlier and severe liver disease. Interferon with ribavirin has become the therapy of choice among people with non-genotype 1a. This is a pilot study to address the relationship of clinical response to combination therapy to the virologic and immunologic parameters. The study will also address the safety and efficacy of the peginterferon alfa-2b among HIV- infected individuals. The predictive ability of baseline HCV viral load, rate of decline of HCV viral load, HIV viral load and CD4 counts to the clinical response of chronic hepatitis to peginterferon and ribavirin will also be studied. Approximately sixty patients who are infected with both HIV and HCV and also have evidence of fibrosis will receive peginterferon alfa-2b and ribavirin for 48 weeks. In order to enroll sixty patients for this study, we will be screening a total of 180 patients. During the 72 weeks study these patients will be monitored for HCV viral load, and other HIV viral load and CD4 counts. Viral kinetics will also be monitored closely and the slope of second, slower phase decline of HCV viral load, which corresponds to the rate of infected cell death presumably may lead to sustained hepatitis C virologic response. The results of the study will enable us to better delineate the possible predictors of sustained response to peginterferon and ribavirin. The safety and tolerability of a combination therapy with peginterferon and ribavirin among HIV-infected individuals on antiretroviral therapy will further define the standard therapy of chronic hepatitis C in HIV-infected individuals.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age greater than or equal to 18 years.

Documentation of HIV-1 infection by any licensed ELISA test and confirmed by a Western Blot.

Documentation of Hepatitis C infection by demonstration of a positive test for hepatitis C antibody.

HCV RNA level greater than 2000 IU/ml by bDNA.

Infected with HCV genotype 1.

Histopathologic features consistent with chronic hepatitis C on liver biopsy at the time of enrollment.

Patients with CD4 greater than 300 cells/mm(3).

Ability to sign informed consent and willingness to comply with the study requirements and clinic policies.

Serum creatinine less than 1.5 mg/dL.

Serum phosphorus greater than or equal to 2.2 mg/dL (normal range NIH 2.3-4.3 mg/dL).

Neutrophil count greater than or equal to 1000 cells/mm(3).

Platelets greater than or equal to 75,000/mm(3).

Hemoglobin greater than or equal to 8.0 mg/dL.

ALT less than 7 times the NIH upper limit of normal.

Serum lipase less than 1.5 times the NIH upper limit of normal.

Not pregnant or breast-feeding. Pregnancy test must be negative within two weeks prior to dosing with study medications.

If capable of pregnancy: use of effective contraception during study: effective contraception methods include abstinence, surgical sterilization of either partner, barrier methods such as diaphragm, condom, cap or sponge, or use of hormonal contraception with an anti-HIV regimen that will not alter metabolism of hormonal contraception. This is advised on the basis of using ribavirin, which may have a potential teratogenic effect in pregnant women.

Need to have a primary doctor outside OP8 who will be taking care of the patients for their HIV infection and liver disease.

Willing to designate a person for durable power of attorney on the NIH form for medical research and medical care purposes at the NIH Clinical Center.

Ability to learn how to safely inject medication subcutaneously.

EXCLUSION CRITERIA:

PT-INR (in the absence of anti-cardiolipin antibody) prolonged by greater than 2 seconds.

Organ transplant recipient.

Elevated alpha-fetoprotein level (greater than 100 ng/mL).

Coexisting neoplastic disease requiring cytotoxic therapy.

Child Pugh's class B.

Severe cardiac or pulmonary decompensation.

Severe liver decompensation or advanced cirrhosis patients.

Severe psychiatric disorder that would interfere with the adherence to protocol requirements.

Preexisting autoimmune disorders including inflammatory bowel diseases, psoriasis, and optic neuritis.

Preexisting uncontrolled seizure disorder.

Severe retinopathy.

Hemoglobinopathy

Direct bilirubin more than or equal to 2 times ULN.

No patients using long term systemic corticosteroids, immunosuppressives, or cytotoxic agents within 60 days of enrollment into the trial.

Chronic viral hepatitis of any other etiology other than hepatitis C.

Active systemic infections other than hepatitis C and HIV.

Liver disease caused by reasons other than hepatitis C like HBV, HDV, Wilson's hemochromatosis, autoimmune hepatitis (ANA greater than 160) except history of drug-associated hepatitis with discontinuation of the causative agent.

Hepatic mass suggestive of hepatocellular carcinoma.

Current alcohol or substance abuse that potentially could interfere with patient compliance.

Significant heart failure.

Evidence of esophageal varices.

Any systemic illness that will make it unlikely that the subject will be able to return to NIH for the required study visits.

Evidence of gastrointestinal malabsorption or chronic nausea or vomiting.

Male partners of pregnant women.

Currently taking didanosine (ddl or Videx-EC or Videx) as part of antiretroviral regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2001-06; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Kottilil, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Result] Rozenberg L, Haagmans BL, Neumann AU, Chen G, McLaughlin M, Levy-Drummer RS, Masur H, Dewar RL, Ferenci P, Silva M, Viola MS, Polis MA, Kottilil S. Therapeutic response to peg-IFN-alpha-2b and ribavirin in HIV/HCV co-infected African-American and Caucasian patients as a function of HCV viral kinetics and interferon pharmacodynamics. AIDS. 2009 Nov 27;23(18):2439-50. doi: 10.1097/QAD.0b013e32832ff1c0. PMID 19898214
- [Result] Avidan NU, Goldstein D, Rozenberg L, McLaughlin M, Ferenci P, Masur H, Buti M, Fauci AS, Polis MA, Kottilil S. Hepatitis C viral kinetics during treatment with peg IFN-alpha-2b in HIV/HCV coinfected patients as a function of baseline CD4+ T-cell counts. J Acquir Immune Defic Syndr. 2009 Dec 1;52(4):452-8. doi: 10.1097/QAI.0b013e3181be7249. PMID 19797971
- [Result] Allison RD, Katsounas A, Koziol DE, Kleiner DE, Alter HJ, Lempicki RA, Wood B, Yang J, Fullmer B, Cortez KJ, Polis MA, Kottilil S. Association of interleukin-15-induced peripheral immune activation with hepatic stellate cell activation in persons coinfected with hepatitis C virus and HIV. J Infect Dis. 2009 Aug 15;200(4):619-23. doi: 10.1086/600107. PMID 19594300
- [Result] Nussenblatt V, McLaughlin M, Rehm CA, Lempicki RA, Brann T, Yang J, Proschan M, Highbarger HC, Dewar RL, Imamichi T, Koratich C, Neumann AU, Masur H, Polis MA, Kottilil S. Immunodeficiency and intrinsic IFN resistance are associated with viral breakthrough to HCV therapy in HIV-coinfected patients. AIDS Res Hum Retroviruses. 2007 Nov;23(11):1354-9. doi: 10.1089/aid.2007.0091. PMID 18184077
- [Result] Neumann A, Polis M, Rozenberg L, Jackson J, Reitano K, McLaughlin M, Koratich C, Dewar R, Masur H, Haagmans B, Kottilil S. Differential antiviral effect of PEG-interferon-alpha-2b on HIV and HCV in the treatment of HIV/HCV co-infected patients. AIDS. 2007 Sep 12;21(14):1855-65. doi: 10.1097/QAD.0b013e32825eaba7. PMID 17721093
- [Result] Wu L, Kottilil S, Lempicki R, Yang J, McLaughlin M, Hu Z, Koratich C, Reitano KN, Rehm CA, Masur H, Wood B, Kleiner DE, Polis MA. Hepatic histologic response (HR) to combination therapy among HCV/HIV-coinfected individuals: interferon induces HR independent of sustained virologic response (SVR). AIDS Res Hum Retroviruses. 2006 Nov;22(11):1091-8. doi: 10.1089/aid.2006.22.1091. PMID 17147494
- [Result] Pau AK, McLaughlin MM, Hu Z, Agyemang AF, Polis MA, Kottilil S. Predictors for hematopoietic growth factors use in HIV/HCV-coinfected patients treated with peginterferon alfa 2b and ribavirin. AIDS Patient Care STDS. 2006 Sep;20(9):612-9. doi: 10.1089/apc.2006.20.612. PMID 16987047
- [Result] Farel C, Suzman DL, McLaughlin M, Campbell C, Koratich C, Masur H, Metcalf JA, Robinson MR, Polis MA, Kottilil S. Serious ophthalmic pathology compromising vision in HCV/HIV co-infected patients treated with peginterferon alpha-2b and ribavirin. AIDS. 2004 Sep 3;18(13):1805-9. doi: 10.1097/00002030-200409030-00009. PMID 15316341
- [Result] Lempicki RA, Polis MA, Yang J, McLaughlin M, Koratich C, Huang DW, Fullmer B, Wu L, Rehm CA, Masur H, Lane HC, Sherman KE, Fauci AS, Kottilil S. Gene expression profiles in hepatitis C virus (HCV) and HIV coinfection: class prediction analyses before treatment predict the outcome of anti-HCV therapy among HIV-coinfected persons. J Infect Dis. 2006 Apr 15;193(8):1172-7. doi: 10.1086/501365. Epub 2006 Mar 13. PMID 16544259
- [Result] Sidique N, Kohli A, Shivakumar B, Migueles S, Subramanian GM, Naggie S, Polis MA, Masur H, Kottilil S. HIV/HCV-coinfected natural viral suppressors have better virologic responses to PEG-IFN and ribavirin than ARV-treated HIV/HCV patients. J Acquir Immune Defic Syndr. 2011 Oct 1;58(2):e38-40. doi: 10.1097/QAI.0b013e31822d463f. No abstract available. PMID 21921725
- [Result] Naggie S, Osinusi A, Katsounas A, Lempicki R, Herrmann E, Thompson AJ, Clark PJ, Patel K, Muir AJ, McHutchison JG, Schlaak JF, Trippler M, Shivakumar B, Masur H, Polis MA, Kottilil S. Dysregulation of innate immunity in hepatitis C virus genotype 1 IL28B-unfavorable genotype patients: impaired viral kinetics and therapeutic response. Hepatology. 2012 Aug;56(2):444-54. doi: 10.1002/hep.25647. Epub 2012 Jul 2. PMID 22331604
- [Result] Osinusi A, Naggie S, Poonia S, Trippler M, Hu Z, Funk E, Schlaak J, Fishbein D, Masur H, Polis M, Kottilil S. ITPA gene polymorphisms significantly affect hemoglobin decline and treatment outcomes in patients coinfected with HIV and HCV. J Med Virol. 2012 Jul;84(7):1106-14. doi: 10.1002/jmv.23302. PMID 22585729
- [Result] Burbelo PD, Kovacs JA, Ching KH, Issa AT, Iadarola MJ, Murphy AA, Schlaak JF, Masur H, Polis MA, Kottilil S. Proteome-wide anti-hepatitis C virus (HCV) and anti-HIV antibody profiling for predicting and monitoring the response to HCV therapy in HIV-coinfected patients. J Infect Dis. 2010 Sep 15;202(6):894-8. doi: 10.1086/655780. PMID 20684729
- [Result] Chary A, Winters MA, Kottilil S, Murphy AA, Polis MA, Holodniy M. Impact of interferon-ribavirin treatment on hepatitis C virus (HCV) protease quasispecies diversity in HIV- and HCV-coinfected patients. J Infect Dis. 2010 Sep 15;202(6):889-93. doi: 10.1086/655784. PMID 20677940

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were all recruited from other NIAID HIV clinical trials and from the nearby Maryland, Virginia and the District of Columbia HIV clinics
Pre-assignment Details: Open label study. The participants were only excluded if they did not meet eligibility criteria, such as pregnancy, availability to make frequent clinic visits and able to meet laboratory safety criteria as described in the clinical protocol.
Groups:
- Peginterferon Alfa-2b, Ribavirin: Weekly Injection (Peginterferon alfa-2b)
  Peginterferon Alfa-2b : Weekly injections for 48 weeks of a dose of 1.5mcg/Kg per week subcutaneously
  Oral Pills (Ribavirin)
  Ribavirin : Weight based Ribavirin dosing 1-1.2grams/day in divided (twice daily) doses for a total duration of 48 weeks.
Period: Overall Study
Arm/Group | Peginterferon Alfa-2b, Ribavirin
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Peg-interefron Alfa 2b, Ribavirin: Weekly Injection
  Peginterferon alpha-2b : Weekly injections for 48 weeks of a dose of 1.5mcg/Kg per week subcutaneously
  Oral Pills
  Ribavirin : Weight based Ribavirin dosing 1-1.2grams/day in divided (twice daily) doses for a total duration of 48 weeks.
Arm/Group | Peg-interefron Alfa 2b, Ribavirin
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 34
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Participants With Viral Decline at Day 3 & 28 With Predictors of Post Treatment Response
Description: HCV viral kinetics were used to predict rates of sustained virology response (SVR) in HIV/HCV connected subjects.
  Measure was determined by analyzing the population of participants with virologic decline of more than 1.0 log at day 3 combined with viral load of less than 5.0 log IU/ml at day 28 to predict sustained virology response
Time Frame: Day 3 and Day 28
Population: Participants with Virologic decline at both Day 3 and absolute HCV VL at Week 28 were analyzed
Measure: Number; unit: participants with post treatment svr
Arm/Group | Peginterferon Alfa-2b, Ribavirin
Number analyzed (Participants) | 23
participants with post treatment svr | 8

ADVERSE EVENTS:
Arm/Group | Peg-interefron Alfa 2b, Ribavirin
Serious Adverse Events (participants affected / at risk) | 3/36
Other Adverse Events (participants affected / at risk) | 20/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peg-interefron Alfa 2b, Ribavirin (N=36)
Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Mild to moderate limitation in activity; some assistance may be needed; no or minimal medical intervention required.
Vision Changes (Eye disorders) | 1 (1) — Transient or mild discomfort; no limitation in activity; no medical intervention/therapy required.
Unusual affect or behavior (Psychiatric disorders) | 1 (1) — Marked limitation in activity; some assistance usually required; medical intervention/therapy required.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peg-interefron Alfa 2b, Ribavirin (N=36)
Anemia (Investigations) | 6 (7) — Hemoglobin decreased
Fatigue (General disorders) | 3 (4)
Neutropenia (Investigations) | 15 (43) — Neutrophil count decreased

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes